CLINICAL TRIAL: NCT01230099
Title: Informing Decisions in Chronic Critical Illness: A Randomized Control Trial (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of North Carolina (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 08-0601 0001 01 ME; R01NR012413-01A1 (NIH)
Record Dates: First submitted 2010-10-22; First posted 2010-10-28 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Critical Illness; Prolonged Mechanical Ventilation
Keywords: Critical Illness; Mechanical Ventilation; Palliative Care; Caregivers
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supportive Information Team Group (Experimental): Protocolized information and support meetings led by palliative care clinicians
  Interventions: Behavioral: Supportive Information Team Group
- Usual Care Group (No Intervention)

INTERVENTIONS:
Behavioral: Supportive Information Team Group — A minimum of two protocolized, interdisciplinary, informational support meetings led by palliative care clinicians will be arranged with family members or other patient surrogates who participate in decision-making for individual chronically critically ill patients.
  Other Names: SIT
  Arms: Supportive Information Team Group

SUMMARY:
The purpose of this study is to test a communication intervention to support family decision-making for patients with chronic critical illness.

DETAILED DESCRIPTION:
Increasing use of intensive care therapies by an aging population has created a new medical syndrome - "chronic critical illness" - encompassing multi-system derangements, recurrent complications, and protracted/permanent dependence on mechanical ventilation and other life-supports. Numbering >100,000 at any point in time, the chronically critically ill are a growing population of older adults and a serious national health problem. Annual expenditures for these patients are estimated at $24 billion, mostly for patients ≥ 65 years old. Yet 6-month mortality rates exceed those for most malignancies, impairments are severe among survivors, and return to the community is rare. Descriptive research has identified domains of information that are important for decision-making by patients/families about continuation of treatment in the chronic phase of critical illness, but has also revealed that decisions are often made without this information or patient goals of care as a context. In acute critical illness, scheduled, structured meetings and printed informational aids are effective for Intensive Care Unit (ICU) families, but no study has tested an intervention to inform and support decision-making about chronic critical illness. This study is a randomized, controlled, multi-center clinical trial of such an intervention. Specific Aims are: (1) To evaluate the impact on family- and patient-focused outcomes of a proactive program of protocolized, interdisciplinary, informational support meetings led by a palliative care physician, plus a printed informational aid, for families of chronically critically ill patients; and (2) To evaluate the impact of this intervention on utilization of critical care resources for the chronically critically ill. We hypothesize that as compared to usual care plus the printed aid, this intervention will effectively inform decision-making, improve family well-being, promote discussion of preferences for patient goals of care, and optimize critical care resource utilization, without increasing patient mortality.

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated ≥ 7 days
* Mechanically ventilated without > 96 hour interruption
* Age ≥ 21 years
* ICU MD does not expect patient will die within 72 hours
* ICU MD does not expect patient will be liberated from the ventilator within 72 hours.

Exclusion Criteria:

* Previous admission to study ICU this hospitalization Mechanically ventilated at outside hospital for > 7 days before transfer
* Chronic Neuromuscular (NM) Disease
* Trauma
* Burn
* Previous palliative care consultation in this hospitalization
* No family or other surrogate decision-maker
* Family not available
* Surrogate lacks English proficiency
* Physician refused permission for research staff to approach the family

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2010-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | Day 90

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Day 18-20
Impact of Events Scale-Revised | Day 90
Discussion of Preferences for Patients Goals of Care | Day 18-20
  Subscale of Center for Gerontology and Health Care Research Toolkit
Quality of Communication | Day 18-20
  Curtis Measure
Family Satisfaction in the Intensive Care Unit (ICU) Survey | Day 90
Modified Center for Gerontology and Health Care Research (CHCR) Tool | Day 90
Limitation of Intensive Care Unit (ICU) Therapy | Average of 60 days
  Percent of patients with mechanical ventilation, renal replacement, vasopressors, or artificial nutrition withheld or withdrawn
Hospital Length of Stay | Average of 60 days
  Days since randomization
Mortality | Day 90
Physician-Surrogate Discordance Score | day 18-20
Discussion of Preferences for Patients Goals of Care | Day 90
  Subscale of Center for Gerontology and Health Care Research Toolkit

CONTACTS AND LOCATIONS:
Overall Officials: Judith Nelson, MD, JD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Shannon Carson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Durham Regional Medical Center, Durham, North Carolina
  - Duke University School of Medicine, Durham, North Carolina

REFERENCES:
- [Derived] Nelson JE, Hanson LC, Keller KL, Carson SS, Cox CE, Tulsky JA, White DB, Chai EJ, Weiss SP, Danis M. The Voice of Surrogate Decision-Makers. Family Responses to Prognostic Information in Chronic Critical Illness. Am J Respir Crit Care Med. 2017 Oct 1;196(7):864-872. doi: 10.1164/rccm.201701-0201OC. PMID 28387538
- [Derived] Carson SS, Cox CE, Wallenstein S, Hanson LC, Danis M, Tulsky JA, Chai E, Nelson JE. Effect of Palliative Care-Led Meetings for Families of Patients With Chronic Critical Illness: A Randomized Clinical Trial. JAMA. 2016 Jul 5;316(1):51-62. doi: 10.1001/jama.2016.8474. Erratum In: JAMA. 2017 May 23;317(20):2134. doi: 10.1001/jama.2017.4298. PMID 27380343